CLINICAL TRIAL: NCT07102238
Title: Lupus Arthritis: Muscoloskeletal Ultrasound as Clinical Outcome of Peripheral Blood and Synovial Deep Phenotyping
Acronym: LUMAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D'Agostino Maria Antonietta, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7740
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLE with muscoloskeletal involvement (Experimental): Consecutive patients with MSK symptoms will be recruited and observed over time. Each enrolled patient will be asked for past and current medical history and treatment. Visits will be scheduled at baseline, at months 3 and 6, then every 6 months up to 18 months, and subsequently according to routine clinical practice. Clinical, laboratory and ultrasound assessments will be conducted at each visit.
  Each patient will be followed for at least 6 months.Important confounding factors such as immune suppression and short/long-term use of NSAIDs at the time of MSK-US will be taken into account. At baseline, a synovial biopsy will be performed at the joint affected by the inflammatory process, and blood samples will be collected.
  Interventions: Procedure: muscoloskeletal ultrasound and synovial biopsy
- other connective tissue diseases with muscoloskeletal involvement (Experimental): Consecutive patients with MSK symptoms will be recruited and observed over time. Each enrolled patient will be asked for past and current medical history and treatment.Clinical, laboratory and ultrasound assessments will be conducted at baseline.
  Important confounding factors such as immune suppression and short/long-term use of NSAIDs at the time of MSK-US will be taken into account.
  At baseline, a synovial biopsy will be performed at the joint affected by the inflammatory process, and blood samples will be collected.
  DAS28, Physician Global Assessment (PGA), Spondylarthritis Research Consortium of Canada (SPARCC) Enthesitis index, Swollen Joint counts (44 or 66) tender joints count (44-66), Widespread Pain Index/Symptom Severity Scale (WPI/SSS) will be collected at each visit. Patients will be treated according to international recommendations and the treating rheumatologist's decision.
  Interventions: Procedure: muscoloskeletal ultrasound and synovial biopsy

INTERVENTIONS:
Procedure: muscoloskeletal ultrasound and synovial biopsy — Use of a standardized US evaluation according with OMERACT definition and scoring system; Synovial biopsy; To identify systemic and synovial disease biomarkers in SLE patients that can predict different joint patterns, systemic manifestations and response to therapy through multi-omics technologies.

SUMMARY:
Musculoskeletal involvement, defined as arthritis/arthralgia, is the most common manifestation of patients with systemic lupus erythematosus (SLE). It accounts for decreased quality of life and can lead to unemployment and disability.

Lupus arthritis is divided into non-erosive, with up to 80% of the cases, erosive, also known as Rhupus, with up to 5% of cases, and deforming, or Jaccoud's arthropathy which can involve up to 15% of the patients. Initially, these 3 forms can present similarly, therefore identifying early on their specific characteristics, can guide better treatments and improve outcomes.

Muscoloskeletal ultrasound (MSK-US) is an established modality to diagnose and investigate joint involvement in inflammatory arthropathies. While for these conditions, well-defined MSK-US approaches exist, much less, if any, for SLE.

The research hypothesis is that a longitudinal standardized prospective MSK-US evaluation coupled with deep phenotyping in patients with SLE peripheral musculoskeletal involvement, will allow us to:

1. better define the systemic nature of this manifestation and
2. yield novel biomarkers that accurately capture this important feature of SLE. In this monocenter study consecutive SLE patients with inflammatory MSK symptoms will recruited and followed prospectively. Patients will undergo MSK ultrasound, blood sample collection, synovial biopsy, for histological assessment. A subgroup of the study cohort will have synovial, Peripheral Blood Mononuclear Cells (PBMCs), serum and omic analysis. Patients will be followed for at least 6 months and up to 18 months with clinical and US evaluation.

Aims and methods

The following two aims are proposed:

1. to define the prevalence and evolution of MSK involvement in SLE patients with inflammatory arthralgia using a standardized US evaluation according with the Outcome Measures in Rheumatology (OMERACT) definition and scoring system In this Aim, a systematic characterization of joint, tendons and enthesis status will be performed through a clinical and US evaluation in order to demonstrate the role of US as an objective tool to better characterize MSK involvement in SLE patients. A MSK-US assessment will be conducted at the beginning and subsequently at each defined time table for all patients.
2. To investigate lupus arthritis with MSK-US, multi-omics technologies including single cell RNA sequencing and proteomics, with the aim to characterize disease activity.

For this Aim, blood and synovial multi-omics analysis will be performed exclusively in a subgroup of 10 SLE recruited patients. A US-guided synovial tissue biopsy will be performed for all patients enrolled in the study, regardless of multi-omics inclusion.

Patients will be longitudinally evaluated to identify clinical articular and systemic flares. The baseline US evaluation and the multi-omics approach will be correlated with the longitudinal manifestations to identify possible biomarkers of flares, both at the joint and systemic levels.

Expected results:

The combined achievement of the above-mentioned aims will address the need to standardize the MSK-US approach and pathogenic mechanisms via biomarkers' discovery of lupus arthritis, a yet still poorly understood SLE manifestation.

expectations:

* To enhance the characterization of joint involvement by reducing the heterogeneity associated with clinical examination through a standardized US evaluation.
* To identify systemic and synovial disease biomarkers in SLE patients that can predict different joint patterns, systemic manifestations and response to therapy through multi-omics technologies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE under ACR/EULAR 2019 criteria [8]
* Age between 18 and 75 years
* Must have inflammatory arthralgia, i.e. signs or symptoms deemed due to active SLE according to the investigator, in relation to distribution and typical inflammatory patterns as previously suggested, including joint symptoms lasting more than 6 weeks, morning stiffness lasting ≥60 minutes, and the most severe symptoms occurring at night and early morning.
* Must be capable of providing informed consent

Exclusion Criteria:

- Patients with contraindications to synovial biopsy or not accepting to perform the synovial biopsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
definition of prevalence of MSK involvement | 18 months
  The percentage of SLE patients with at least one joint, tendon or enthesis showing signs of inflammation (synovitis, tenosynovitis, enthesitis) detected by musculoskeletal ultrasound (MSK-US) using OMERACT definitions and EULAR-OMERACT scoring systems.

SECONDARY OUTCOMES:
Identification of candidate biomarkers associated with MSK disease activity and flares in SLE | 18 months
  Number of transcripts (from single-cell RNA sequencing of PBMCs and spatial transcriptomics of synovial tissue) and proteins (from Olink proteomic assay in plasma) significantly associated with MSK-US findings and systemic disease flares over the 18-month follow-up. Associations will be evaluated using differential expression analysis and Gene Association with Multiple Traits (GAMuT) statistical models.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonietta D'Agostino, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No